CLINICAL TRIAL: NCT05042102
Title: The Combination of Donepezil and Cognitive Training for Treating Alcohol Use Disorder
Brief Title: Donepezil and Cognitive Training for Alcohol Use Disorder (AUD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Yale University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GY0010; 5R01AA029075 (NIH)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Donepezil + Cognitive remediation therapy (CRT) (Experimental): Subjects in this arm will receive (1) donepezil and (2) cognitive remediation therapy (CRT). Subjects will take 5 mg/day of oral donepezil in the evening for the first 4 weeks, then 10 mg/day of oral donepezil in the evening until week 13.
  Interventions: Combination Product: Donepezil + Cognitive remediation therapy (CRT)
- Donepezil + Placebo CRT (Experimental): Subjects in this arm will receive (1) donepezil and (2) placebo CRT. Subjects will take 5 mg/day of oral donepezil in the evening for the first 4 weeks, then 10 mg/day of oral donepezil in the evening until week 13.
  Interventions: Combination Product: Donepezil + Placebo CRT
- Placebo medication + Cognitive remediation therapy (CRT) (Experimental): Subjects in this arm will receive (1) placebo medication and (2) cognitive remediation therapy (CRT). Subjects will take placebo oral medication in the evening for the first 4 weeks, then placebo oral medication in the evening until week 13.
  Interventions: Combination Product: Placebo medication + Cognitive remediation therapy (CRT)
- Placebo medication + Placebo CRT (Experimental): Subjects in this arm will receive (1) placebo medication and (2) placebo CRT. Subjects will take placebo oral medication in the evening for the first 4 weeks, then placebo oral medication in the evening until week 13.
  Interventions: Combination Product: Placebo medication + Placebo CRT

INTERVENTIONS:
Combination Product: Donepezil + Cognitive remediation therapy (CRT) — Subjects in this arm will receive (1) donepezil and (2) cognitive remediation therapy (CRT). Subjects will take 5 mg/day of oral donepezil in the evening for the first 4 weeks, then 10 mg/day of oral donepezil in the evening until week 13.
  Arms: Donepezil + Cognitive remediation therapy (CRT)
Combination Product: Donepezil + Placebo CRT — Subjects in this arm will receive (1) donepezil and (2) placebo CRT. Subjects will take 5 mg/day of oral donepezil in the evening for the first 4 weeks, then 10 mg/day of oral donepezil in the evening until week 13.
  Arms: Donepezil + Placebo CRT
Combination Product: Placebo medication + Cognitive remediation therapy (CRT) — Subjects in this arm will receive (1) placebo medication and (2) cognitive remediation therapy (CRT). Subjects will take placebo oral medication in the evening for the first 4 weeks, then placebo oral medication in the evening until week 13.
  Arms: Placebo medication + Cognitive remediation therapy (CRT)
Combination Product: Placebo medication + Placebo CRT — Subjects in this arm will receive (1) placebo medication and (2) placebo CRT. Subjects will take placebo oral medication in the evening for the first 4 weeks, then placebo oral medication in the evening until week 13.
  Arms: Placebo medication + Placebo CRT

SUMMARY:
The goal of the project is to evaluate whether donepezil + cognitive remediation therapy is superior to placebo in reducing heavy drinking in patients with alcohol use disorder in a double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion criteria:

1. Males and females 18-80 years of age
2. Fluency in English and a 6th grade or higher reading level
3. Meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a current alcohol use disorder (subjects should have a primary alcohol use disorder [AUD] diagnosis, but may have concurrent occasional use of other substances)
4. Last alcohol use and at least one heavy drinking day within the past 30 days
5. Willingness to attend follow-up assessments at 13 weeks
6. Willingness to submit to Urine Toxicology screenings

Exclusion criteria:

1. Lifetime diagnosis of a psychotic disorder, not induced by drug use
2. Current treatment with opioids or benzodiazepines, which may affect new learning
3. Involvement in a legal case that may lead to incarceration during the study period
4. Residential plans that would interfere with participation
5. Medical illness that may significantly compromise cognition (e.g., Parkinson's, Alzheimer's, Huntington's chorea, moderate or greater TBI)
6. An uncorrected sensory impairment (hearing or sight) that would seriously interfere with cognitive training
7. Pre-morbid intelligence quotient (IQ) estimate below 70
8. Unstable housing or lack of commitment to staying within a geographic area that would make follow-up unlikely
9. Unwillingness to provide contact information of someone who can help study staff contact the subjects in the event that study staff are unable to maintain contact directly
10. Allergy to donepezil
11. Unstable cardiovascular disease or unstable medical condition-clinically determined by a physician
12. Imminent suicidal or homicidal risk
13. Pregnant or nursing women, positive pregnancy test, or inadequate birth control methods in women of childbearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Heavy drinking days | 13 weeks of active intervention
  Heavy drinking days as measured by weekly Time Line Follow Back (TLFB)

SECONDARY OUTCOMES:
Global neurocognitive functioning | At 7 weeks and at 13 weeks
  Global neurocognitive functioning on a global index of neurocognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Gihyun Yoon, MD, Principal Investigator — Yale University, VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yoon G, Sofuoglu M, Petrakis IL, Pittman B, Bell MD. The combination of donepezil and cognitive training for improving treatment outcomes for alcohol use disorder: Design of a randomized controlled trial. Contemp Clin Trials. 2024 Oct;145:107657. doi: 10.1016/j.cct.2024.107657. Epub 2024 Aug 5. PMID 39111388